CLINICAL TRIAL: NCT04906421
Title: A Phase 2B, Multi-Center, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of TVB-2640 in Subjects With Nonalcoholic Steatohepatitis (FASCINATE-2)
Brief Title: Study of TVB-2640 in Subjects With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB2640-CLIN-007
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Dysfunction-assocated Steatohepatitis/ Nonalcoholic Fatty Liver Disease
Keywords: NASH; Nonalcoholic Steatohepatitis; Fatty Liver Disease; Biopsy Confirmed; FASN; Fatty Liver; Liver Disease; Digestive System Diseases; MASH; Metabolic dysfunction-associated steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases; Digestive System Diseases | interventions — TVB-2640

STUDY DESIGN:
Intervention Model Description: Subjects with liver fibrosis stage F2-F3, will be enrolled and randomized in a 2:1 ratio to receive TVB-2640, or placebo PO QD
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TVB-2640 50 mg (Experimental): Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  Interventions: Drug: TVB-2640
- Placebo (Placebo Comparator): Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TVB-2640 — Oral dose, tablet
  Arms: TVB-2640 50 mg
Other: Placebo — Oral dose, tablet
  Arms: Placebo

SUMMARY:
This is a Phase 2, multi-center, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy on TVB-2640 in subjects with non-alcoholic steatohepatitis (NASH). Subjects will be randomly assigned toTVB-2640 or matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.

DETAILED DESCRIPTION:
The indication nonalcoholic steatohepatitis [NASH]) is now referred to as metabolic dysfunction-associated steatohepatitis (MASH) and is characterized by hepatocyte necrosis, chronic inflammation, and resultant fibrosis formation.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to participate in the study and provide written informed consent.
* Male and female adults ≥18 years of age on the date that written informed consent to take part in the study is provided.
* Body mass index (BMI) ≥23 kg/m2 for Asians and ≥25 kg/m2 for other races.
* Female subjects must be either:

  * Not of childbearing potential OR
  * Women of childbearing potential (WOCBP) must have a negative serum pregnancy (beta-human chorionic gonadotropin [β-HCG]) test during Screening, a negative urine pregnancy test within 24 hours before the first dose of study drug on Day 1, and must agree to perform urine home pregnancy tests monthly between study visits. WOCBP must not be breastfeeding, not plan to become pregnant during the study, and must use birth control.
* Must have liver stiffness measurement ≥8.5 kPa measured by FibroScan and CAP score measured by FibroScan ≥280 dB/m during the Screening period.
* Histologic confirmation of NASH: must have had prior liver biopsy within 180 days before randomization (randomization is within 24 hours of Baseline [Day1]) with fibrosis stage F2-F3 and a NAS of ≥4 with at least a score of 1 in each of the following NAS components: steatosis, ballooning degeneration, and lobular inflammation.

Exclusion Criteria:

* History of harmful alcohol intake for a period of more than 3 consecutive months within 1 year prior to Screening in the judgement of the Investigator.
* Active substance abuse.
* Gain or loss of >5% of body weight in the 6 months prior to Baseline (Day 1) or >10% of body weight in the 12 months prior to Screening.
* Type 1 diabetes mellitus by history.
* Positive severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) polymerase chain reaction (PCR) test within 30 days before Baseline, history of hospitalization for coronavirus disease-2019 (COVID-19) ), or history of use of oxygen due to COVID-19) <6 months prior to the Screening visit date. Note that previous COVID-19 infection alone is not exclusionary and vaccination against SARS-CoV-2 is allowed. Infection and/or vaccination must be documented.
* Uncontrolled T2DM, defined as HbA1c ≥9.5% at Screening.
* Presence of cirrhosis on liver histology (stage 4 fibrosis), according to the judgement of the central reader, and/or cross sectional imaging evidence consistent with cirrhosis and/or portal hypertension.
* Use of glucagon-like peptide-1 (GLP-1) agonists or a sodium-glucose co-transporter-2 (SGLT2) inhibitor, unless on a stable daily dose for at least 6 months prior to the Screening visit date, or on a complex oral anti-diabetic (OAD) regimen (3 or more OADs [except for a GLP-1 agonist or an SGLT2 inhibitor]), unless on a stable dose for at least 3 months prior to the Screening visit date.
* Subjects with active or quiescent chronic liver disease of etiologies other than NASH (eg, viral or autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cholangitis, and 'autoimmune hepatitis-overlap' syndromes, hemochromatosis, Wilson's disease, alpha 1 antitrypsin deficiency, alcohol-related liver disease, drug-induced liver disease, and/or infiltrative conditions [eg, sarcoidosis]).
* Current or historic clinically evident hepatic decompensation event (eg, ascites formation, variceal hemorrhage, hepatic encephalopathy).
* Any subject who has sustained a clinically evident cardiovascular, cerebrovascular, and/or peripheral vascular event during the 12 months prior to anticipated Baseline (Day 1) visit date is not eligible for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (117):
- United States (103):
  - North Alabama Health Research, Huntsville, Alabama
  - North Alabama GI Research Center, Madison, Alabama
  - GI Alliance Arizona Digestive Health-Sun City, Sun City, Arizona
  - ARcare Center for Clinical Research, LLC - Conway, Conway, Arkansas
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - Liver Wellness Center, Little Rock, Arkansas
  - Citrus Valley Gastroenterology, Covina, California
  - UCSD, NAFLD Research Center / Altman Clinical and Translational Research Institute, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Clinical Trials Research, Lincoln, California
  - Digestive Health Research of Southern California LLC, Long Beach, California
  - Digestive Health Research of Southern California, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - United Medical Doctors, Murrieta, California
  - Palmtree Clinical Research, INC, Palm Springs, California
  - IVGI, Ventura, California
  - Gastro Florida, Clearwater, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - American Research Institute, Inc, Cutler Bay, Florida
  - Top Medical Research, Inc, Cutler Bay, Florida
  - Covenant Metabolic Specialists, LLC, Fort Myers, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Miguel A Rebollar, MD PA, Hialeah, Florida
  - Global Research Associates, Homestead, Florida
  - Ocala GI Research dba Lake Center for Clinical Research, LLC, Lady Lake, Florida
  - Accel Research Site - Maitland, Maitland, Florida
  - CPMI, Miami, Florida
  - University of Miami, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Genoma Research Group, Inc, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Professional Medical Research, Miramar, Florida
  - Ocala GI Research, LLC, Ocala, Florida
  - Innovation Medical Research Center, Inc, Palmetto Bay, Florida
  - Pensacola GI Research Center, LLC, Pensacola, Florida
  - Covenant Metabolic Specialists, LLC, Sarasota, Florida
  - Headlands Research Sarasota, Sarasota, Florida
  - Conquest Research, Winter Park, Florida
  - Summit Clinical Research, Athens, Georgia
  - Southeast Clinical Research Center, Dalton, Georgia
  - Care Access Research, Fairview Heights, Illinois
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Greater Boston Gastroenterology, Boston, Massachusetts
  - Greater Boston Gastroenterology, Framingham, Massachusetts
  - FC Research LLC, South Dartmouth, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - GI Associates Research, LLC, Columbia, Missouri
  - Sierra Clinical Research, Las Vegas, Nevada
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Care Access, Yonkers, New York
  - University of North Carolina at Chapel Hill. UNC Liver Center, Chapel Hill, North Carolina
  - Northeast GI Research Division, Concord, North Carolina
  - ACME Medical Specialties PLCC, Lumberton, North Carolina
  - Care Access Research, Lumberton, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Ohio State University, Columbus, Ohio
  - DSI Research, LLC - Northridge, Dayton, Ohio
  - Care Access Research, Poland, Ohio
  - DDSI Clinical Trials, Oklahoma City, Oklahoma
  - University of Gastroenterology, Providence, Rhode Island
  - Care Access Research, Warwick, Rhode Island
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Columbia Digestive Health Research, LLC, Columbia, South Carolina
  - Digestive Disease Research Center LLC, Greenwood, South Carolina
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Cordova, Tennessee
  - Gastro One, Germantown, Tennessee
  - Digestive Health Research, Lebanon, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - Apex Mobile Clinical Research, LLC, Bellaire, Texas
  - Texas Digestive Disease Consultants - Cedar Park, Cedar Park, Texas
  - The Liver Institute at Methodist Health System, Dallas, Texas
  - GI Alliance -Texas Digestive Disease Consultants, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Texas Digestive Disease Consultants - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - GI Alliance / Texas Digestive Disease Consultants, Lubbock, Texas
  - Centex Studies, McAllen, Texas
  - ClinRx Research LLC, Plano, Texas
  - American Research Corporation, San Antonio, Texas
  - Clinical Trials of Texas Inc., San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Impact Research Institute, Waco, Texas
  - Digestive Health Research of North Texas, Wichita Falls, Texas
  - Care Access, Ogden, Utah
  - Bon Secours Richmond Community Hospital LLC d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - GI Select Health Research, LLC, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Gastroenterology Consultants of SW Virginia, Roanoke, Virginia
- Canada (6):
  - University of Calgary Liver Unit, Calgary, Alberta
  - GI Research Institute, Vancouver, British Columbia
  - Office of Dr. Gauthier, North Bay, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Office of Dr. Gauthier, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Poland (7):
  - Centrum Medyczne Pratia, Katowice
  - Krakowskie Centrum Medyczne sp z o.o., Krakow
  - Hepatology Outpatient Clinic, Śląskie
  - ID Clinic Arkadiusz Pisula, Śląskie
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Medyczne K2J2, Wołomin
  - FutureMeds, Wroclaw
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loomba R, Bedossa P, Grimmer K, Kemble G, Bruno Martins E, McCulloch W, O'Farrell M, Tsai WW, Cobiella J, Lawitz E, Rudraraju M, Harrison SA. Denifanstat for the treatment of metabolic dysfunction-associated steatohepatitis: a multicentre, double-blind, randomised, placebo-controlled, phase 2b trial. Lancet Gastroenterol Hepatol. 2024 Dec;9(12):1090-1100. doi: 10.1016/S2468-1253(24)00246-2. Epub 2024 Oct 11. PMID 39396529
- See also: Denifanstat for the treatment of metabolic dysfunctionassociated steatohepatitis: a multicentre, double-blind, randomised, placebo-controlled, phase 2b trial — https://pubmed.ncbi.nlm.nih.gov/39396529/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TVB-2640 50 mg | Placebo
Started | 112 | 56
mITT | 81 | 45
Completed | 80 | 47
Not Completed | 32 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TVB-2640 50 mg | Placebo | Total
Number analyzed (Participants) | 112 | 56 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.5) | 58.4 (11.9) | 57.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 34 | 100
  Male | 46 | 22 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 21 | 55
  Not Hispanic or Latino | 78 | 35 | 113
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 4 | 11
  White | 100 | 50 | 150
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Histological Improvement in Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) Without Worsening of Fibrosis (by NASH Clinical Research Network [CRN] Fibrosis Score).
Description: Histological improvement is defined as ≥2 points improvement in NAS with ≥1 point improvement in ballooning or inflammation
Time Frame: 52 Weeks
Population: ITT and mITT Population
Measure: Count of Participants; unit: Participants
Groups:
- ITT: TVB-2640 50 mg: Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  TVB-2640: Oral dose, tablet
- ITT: Placebo: Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Placebo: Oral dose, tablet
- mITT: TVB-2640 50 mg: Comprises all subjects in the ITT population who have completed at least 42 weeks of treatment and have an evaluable post treatment histological assessment.
  TVB-2640: Oral dose, tablet
- mITT: Placebo: Comprises all subjects in the ITT population who have completed at least 42 weeks of treatment and have an evaluable post treatment histological assessment.
  Placebo: Oral dose, tablet
Arm/Group | ITT: TVB-2640 50 mg | ITT: Placebo | mITT: TVB-2640 50 mg | mITT: Placebo
Number analyzed (Participants) | 112 | 56 | 81 | 45
Participants | 42 | 9 | 42 | 9
Statistical Analysis 1: Comparison: ITT: TVB-2640 50 mg vs ITT: Placebo; ITT Population analysis; Test type: Superiority; p = 0.0018, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); One-sided
Statistical Analysis 2: Comparison: ITT: TVB-2640 50 mg vs ITT: Placebo; ITT Population Analysis; Test type: Superiority; p = 0.0035, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided
Statistical Analysis 3: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0001, t-test, 1 sided — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); One-sided
Statistical Analysis 4: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided

2. Primary Outcome: Subjects With Resolution of Steatohepatitis and No Worsening of Liver Fibrosis by NASH CRN Fibrosis Score and Histological Improvement in NAS.
Description: NASH resolution defined as absence of fatty liver disease or isolated or simple steatosis without steatohepatitis and a score of either 0 or 1 for inflammation, 0 for ballooning and any value for steatosis and no worsening of liver fibrosis (by NASH CRN fibrosis score). Histological improvement defined as ≥2 point improvement in NAS (with ≥1 point improvement in ballooning or inflammation).
Time Frame: 52 Weeks
Population: ITT and mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | ITT: TVB-2640 50 mg | ITT: Placebo | mITT: TVB-2640 50 mg | mITT: Placebo
Number analyzed (Participants) | 112 | 56 | 81 | 45
Participants | 29 | 6 | 29 | 6
Statistical Analysis 1: Comparison: ITT: TVB-2640 50 mg vs ITT: Placebo; ITT Population Analysis; Test type: Superiority; p = 0.0087, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); One-sided
Statistical Analysis 2: Comparison: ITT: TVB-2640 50 mg vs ITT: Placebo; ITT Population Analysis; Test type: Superiority; p = 0.0173, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided
Statistical Analysis 3: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); One-sided
Statistical Analysis 4: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0044, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided

3. Secondary Outcome: Proportion of Subjects Experiencing Fibrosis Improvement of ≥1 Stage by NASH CRN Score Without Worsening of Steatohepatitis
Description: Proportion of subjects experiencing fibrosis improvement of ≥1 stage by NASH CRN score Without worsening of steatohepatitis (defined as no increase in NAS for ballooning, inflammation, or steatosis) at 52 weeks.
Time Frame: 52 Weeks
Population: mITT Population and Subgroups
Measure: Count of Participants; unit: Participants
Groups:
- mITT: TVB-2640 50 mg: Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  Comprises all subjects in the ITT population who have completed at least 42 weeks of treatment and have an evaluable post treatment histological assessment.
  TVB-2640: Oral dose, tablet
- mITT: Placebo: Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Comprises all subjects in the ITT population who have completed at least 42 weeks of treatment and have an evaluable post treatment histological assessment.
  Placebo: Oral dose, tablet
- Subgroup: Fibrosis Stage F2; TVB-2640: Subgroup of Fibrosis Stage F2 at Baseline
  Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  TVB-2640: Oral dose, tablet
- Subgroup: Fibrosis Stage F2; Placebo: Subgroup: Fibrosis Stage F2 at Baseline
  Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Placebo: Oral dose, tablet
- Subgroup: Fibrosis Stage F3; TVB-2640: Subgroup of Fibrosis Stage F3 at Baseline
  Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  TVB-2640: Oral dose, tablet
- Subgroup: Fibrosis Stage F3; Placebo: Subgroup: Fibrosis Stage F3 at Baseline
  Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Placebo: Oral dose, tablet
- Subgroup: T2DM; TVB-2640: Subgroup of Type 2 Diabetes Mellitus at Baseline
  Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  TVB-2640: Oral dose, tablet
- Subgroup: T2DM; Placebo: Subgroup: Type 2 Diabetes Mellitus at Baseline
  Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Placebo: Oral dose, tablet
Arm/Group | mITT: TVB-2640 50 mg | mITT: Placebo | Subgroup: Fibrosis Stage F2; TVB-2640 | Subgroup: Fibrosis Stage F2; Placebo | Subgroup: Fibrosis Stage F3; TVB-2640 | Subgroup: Fibrosis Stage F3; Placebo | Subgroup: T2DM; TVB-2640 | Subgroup: T2DM; Placebo
Number analyzed (Participants) | 81 | 45 | 34 | 22 | 47 | 23 | 55 | 27
Participants | 33 | 8 | 10 | 5 | 23 | 3 | 22 | 5
Statistical Analysis 1: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0102, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided
Statistical Analysis 2: Comparison: Subgroup: Fibrosis Stage F2; TVB-2640 vs Subgroup: Fibrosis Stage F2; Placebo; Subgroup Fibrosis Stage F2 at Baseline Population Analysis; Test type: Superiority; p = 0.59, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided
Statistical Analysis 3: Comparison: Subgroup: Fibrosis Stage F3; TVB-2640 vs Subgroup: Fibrosis Stage F3; Placebo; Subgroup Fibrosis Stage F3 at Baseline Population Analysis; Test type: Superiority; p = 0.0032, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-Sided
Statistical Analysis 4: Comparison: Subgroup: T2DM; TVB-2640 vs Subgroup: T2DM; Placebo; Subgroup Type 2 Diabetes Mellitus at Baseline Population Analysis; Test type: Superiority; p = 0.0764, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided

4. Secondary Outcome: Proportion of Subjects Experiencing Resolution of Steatohepatitis and no Worsening of Liver Fibrosis (by NASH CRN Fibrosis Score)
Description: Resolution of steatohepatitis is defined as absence of fatty liver disease or isolated or simple steatosis without steatohepatitis and a NAS of 0 or 1 for inflammation, 0 for ballooning, and any value for steatosis.
Time Frame: 52 Weeks
Population: mITT Population
Measure: Count of Participants; unit: Participants
Groups:
- mITT: TVB-2640 50 mg: Subjects will receive TVB-2640 PO QD for 52 weeks, with the first dose administered on Day 1.
  TVB-2640: Oral dose, tablet
- mITT: Placebo: Subjects will receive matching placebo PO QD for 52 weeks, with the first dose administered on Day 1.
  Placebo: Oral dose, tablet
Arm/Group | mITT: TVB-2640 50 mg | mITT: Placebo
Number analyzed (Participants) | 81 | 45
Participants | 31 | 7
Statistical Analysis 1: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0043, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided

5. Secondary Outcome: Proportion of Subjects With Improvement in Liver Fibrosis >=1 Stage by NASH CRN Fibrosis Score Without Worsening of Steatohepatitis at 52 Weeks OR Resolution of Steatohepatitis and No Worsening of Liver Fibrosis by NASH CRN Fibrosis Score
Description: No increase in NAS for ballooning, inflammation or steatosis.
Time Frame: 52 Weeks
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | mITT: TVB-2640 50 mg | mITT: Placebo
Number analyzed (Participants) | 81 | 45
Participants | 45 | 12
Statistical Analysis 1: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p = 0.0018, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided

6. Secondary Outcome: Proportion of MRI-PDFF ≥30% Responders.
Description: MRI PDFF ≥30% responder is defined as a subject with ≥8% liver fat content at Baseline who achieves a relative reduction from Baseline in MRI-PDFF ≥30%.
Time Frame: 52 Weeks
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | mITT: TVB-2640 50 mg | mITT: Placebo
Number analyzed (Participants) | 81 | 45
Participants | 69 | 38
Statistical Analysis 1: Comparison: mITT: TVB-2640 50 mg vs mITT: Placebo; mITT Population Analysis; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified CMH test stratified by T2DM status at baseline (yes or no) and amount of fibrosis at baseline (F2 or F3); Two-sided

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | TVB-2640 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/56
Serious Adverse Events (participants affected / at risk) | 13/112 | 3/56
Other Adverse Events (participants affected / at risk) | 79/112 | 36/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TVB-2640 50 mg (N=112) | Placebo (N=56)
Cellulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Norovirus infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Bell's palsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 0 | 1
Bronchoscopy (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TVB-2640 50 mg (N=112) | Placebo (N=56)
COVID-19 (Infections and infestations) | 19 | 6
Urinary tract infection (Infections and infestations) | 9 | 3
Sinusitis (Infections and infestations) | 6 | 2
Dry Eye (Eye disorders) | 10 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 5 | 3
Headache (Nervous system disorders) | 5 | 3
Depression (Psychiatric disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT04906421/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT04906421/SAP_001.pdf